CLINICAL TRIAL: NCT02136459
Title: Assessment of Non-neural Voice Changes in Thyroidectomy Patients: A Randomized Control Trial
Brief Title: Non-neural Vocal Changes After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Infirmary-Victoria University Hospital (Other)
Responsible Party: Principal Investigator, Patrick Sheahan, Consultant Otolaryngologist Head and neck Surgeon, South Infirmary-Victoria University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIVUH1
Record Dates: First submitted 2014-05-06; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Thyroidectomy
Keywords: Thyroidectomy; Endotracheal tube; Voice; Complications; Patients undergoing elective thyroidectomy
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small tube size (Experimental): Size 6.5 ETT for female, size 7.0 ETT for male
  Interventions: Other: Small Tube size
- Large tube size (Active Comparator): Normal tube size, size 7.5 for female, size 8 for male
  Interventions: Other: Large Tube size

INTERVENTIONS:
Other: Small Tube size — An endotracheal tube of size 6.5 in females and 7.0 in males was used for endotracheal intubation of patients undergoing thyroid surgery
  Other Names: Smaller size of endotracheal tube (ETT) inserted
  Arms: Small tube size
Other: Large Tube size — An endotracheal tube of size 7.5 in females and 8.0 in males was used for endotracheal intubation of patients undergoing thyroid surgery
  Other Names: Standard size endotracheal tube
  Arms: Large tube size

SUMMARY:
The purpose of this study is to test the investigators hypothesis that intubation with a smaller ETT would lead to reduced postoperative vocal impairment and laryngoscopic evidence of laryngeal trauma than intubation with a standard size ETT.

DETAILED DESCRIPTION:
The optimum size of endotracheal tube (ETT) for general anaesthesia remains a matter of debate. Choice of ETT size may be of particular pertinence during thyroid surgery, for a number or reasons. Because of the strong attachments of the thyroid gland to the trachea, intraoperative mobilization of the thyroid will lead to inevitable movement of the trachea and larynx against the fixed ETT, with consequent risk of traumatic injury to tracheal mucosa, vocal cords, and arytenoids. Thus thyroidectomy is likely to be associated with a greater risk of laryngeal trauma related to the ETT than operations outside the Head and Neck region where there is no movement of the larynx. On top of this, postoperative vocal impairment comprises one of the most important concerns after thyroidectomy, usually attributed to impaired vocal fold function secondary to recurrent laryngeal nerve injury. However, post-thyroidectomy vocal impairment can also occur in cases where the recurrent laryngeal nerve is preserved. Thus, concerns regarding vocal outcomes after thyroidectomy tend to be foremost in the mind of both the surgeon and the patient, and any measures which can be taken to minimize post-thyroidectomy hoarseness, which might include choosing the optimal ETT size, would appear to constitute a worthwhile endeavor.

Laryngeal trauma due to endotracheal intubation is probably more common than appreciated, however, given that symptoms of sore throat and hoarseness after most operations are generally self-limiting, this is not usually a major cause of concern. On the other hand, postoperative vocal symptoms may be a major cause of anxiety after thyroidectomy, due to fear of damage to the recurrent laryngeal nerve or the external branch of the superior laryngeal nerve (SLN). Laryngeal trauma without impairment of vocal fold function has been reported to be a significant cause of vocal symptoms after thyroid surgery. However, no previously published study has attempted to correlate post-thyroidectomy vocal symptoms or signs of laryngeal trauma with ETT size.

The hypothesis of the present study was that intubation with a smaller size ETT would lead to less trauma to the larynx during thyroidectomy than intubation with a standard size tube, and this would be reflected through less postoperative throat symptoms and objective laryngeal alterations. The rationale for this hypothesis was that a smaller caliber tube would be less unyielding when the larynx is moved against it, and thus would lead to less laryngeal injury. In order to address this question, the investigators designed a randomized controlled trial, comparing the impact of intubation with a smaller size tube (size 6.5 for females, and size 7 for males) with that of intubation with ETTs of the standard size used in the investigators department (size 7.5 for females, and size 8 for males).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and over scheduled to undergo thyroid surgery performed by one of two surgeons for benign or malignant thyroid disease during the study

Exclusion Criteria:

* pre-existing vocal cord palsy or major vocal cord pathology; patients with invasive thyroid cancers; and patients undergoing concomitant lateral neck dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Laryngoscopic appearance | 24 hours
  A laryngoscopic score of 0,1,2 was given according to absence (0), presence (1) or presence of severe (2) findings of each the following laryngoscopic findings: erythema, oedema, polyp or nodule, and reduced vocal mobility

SECONDARY OUTCOMES:
Vocal outcomes | 24 hours
  Grade, roughness, breathiness, aesthenia and strain (GRBAS) score
Laryngoscopic appearance | 3 weeks
  A laryngoscopic score of 0,1,2 was given according to absence (0), presence (1) or presence of severe (2) findings of each the following laryngoscopic findings: erythema, oedema, polyp or nodule, and reduced vocal mobility
Objective vocal outcomes | 3 weeks
  Grade, roughness, breathiness, aesthenia and strain (GRBAS) score
Subjective vocal outcomes | 3 weeks
  VHI (Voice Handicap Index) scores

OTHER OUTCOMES:
Pain | 24 hours
  VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Rania Mehanna, Principal Investigator — South Infirmary-Victoria University Hospital
Locations (1):
- South Infirmary Victoria University Hospital, Cork, Ireland

REFERENCES:
- [Derived] Mehanna R, Hennessy A, Mannion S, O'Leary G, Sheahan P. Effect of Endotracheal Tube Size on Vocal Outcomes After Thyroidectomy: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Aug;141(8):690-5. doi: 10.1001/jamaoto.2015.1198. PMID 26158868